CLINICAL TRIAL: NCT04368585
Title: An Open-Label, 3-Period, Fixed-Sequence, Study to Examine the Effect of Aluminum Hydroxide/Magnesium Hydroxide/Simethicone and Omeprazole on the Single-Dose Pharmacokinetics of Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) in Healthy Adult Subjects
Brief Title: Study to Examine the Effect of Antacid and Omeprazole on the Single-Dose Pharmacokinetics of Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPR994-107
Record Dates: First submitted 2020-04-09; First posted 2020-04-30 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tebipenem; Aluminum Hydroxide; Magnesium Hydroxide; Simethicone; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TBPM-PI-HBr Alone (Period 1) (Experimental): Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) 600 mg single-dose given orally alone.
  Interventions: Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr)
- TBPM-PI-HBr and Antacid (Period 2) (Experimental): 20 mL aluminum hydroxide/magnesium hydroxide/simethicone (400 mg aluminum hydroxide/400 mg magnesium hydroxide/40 mg simethicone per 5 mL) oral suspension will be coadministered with 600 mg (2 x 300 mg tablets) TBPM-PI-HBr at Hour 0 on Day 1.
  Interventions: Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr); Drug: 20 mL aluminum hydroxide/magnesium hydroxide/simethicone (400 mg aluminum hydroxide/400 mg magnesium hydroxide/40 mg simethicone per 5 mL)
- TBPM-PI-HBr and Omeprazole (Period 3) (Experimental): 40 mg (1 x 40 mg capsule) omeprazole administered QD at Hour -2 on Days 1 through 5, with 600 mg (2 x 300 mg tablets) TBPM-PI-HBr administered at Hour 0 on Day 5.
  Interventions: Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr); Drug: Omeprazole

INTERVENTIONS:
Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) — Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) 600 mg single-dose given orally.
  Other Names: TBPM-PI-HBr; SPR994
Drug: 20 mL aluminum hydroxide/magnesium hydroxide/simethicone (400 mg aluminum hydroxide/400 mg magnesium hydroxide/40 mg simethicone per 5 mL) — 20 mL aluminum hydroxide/magnesium hydroxide/simethicone (400 mg aluminum hydroxide/400 mg magnesium hydroxide/40 mg simethicone per 5 mL) oral suspension.
  Arms: TBPM-PI-HBr and Antacid (Period 2)
Drug: Omeprazole — 40 mg (1 x 40 mg capsule) omeprazole administered QD
  Arms: TBPM-PI-HBr and Omeprazole (Period 3)

SUMMARY:
To assess the effect of a single dose of aluminum hydroxide/magnesium hydroxide/simethicone and omeprazole on the pharmacokinetics (PK) of TBPM, following a single dose of TBPM-PI-HBr in healthy adult subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy, adult, male or female, 18-55 years of age, inclusive, at the screening visit.
* Continuous non-smoker
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at the screening visit.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.

Key Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected to have during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* History of significant allergic disease requiring treatment
* History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds (especially fluoroquinolone-, carbapenem-, penicillin-, and cephalosporin-antibiotics sensitivity).
* History of known genetic metabolism anomaly associated with carnitine deficiency (e.g., carnitine transporter defect, methylmalonic aciduria, propionic acidemia).
* History of cholecystectomy.
* Female subjects with a positive pregnancy test at the screening visit or first check-in or who are lactating.
* Positive urine drug or alcohol results at the screening visit or first check-in.
* Positive results at the screening visit for human immunodeficiency virus (HIV 1 and 2), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve, from time 0 to the last observed non-zero concentration (t). | Day 2 (Periods 1 and 2) and Day 6 (Period 3)
Area under the curve extrapolated to infinity (AUC0-∞). | Day 2 (Periods 1 and 2) and Day 6 (Period 3)
Percent of AUC0-inf extrapolated (AUC%extrap) | Day 2 (Periods 1 and 2) and Day 6 (Period 3)
Maximum plasma concentration (Cmax). | Day 2 (Periods 1 and 2) and Day 6 (Period 3)
Time to the maximum plasma concentration (Tmax). | Day 2 (Periods 1 and 2) and Day 6 (Period 3)
Terminal elimination half-life (t½). | Day 2 (Periods 1 and 2) and Day 6 (Period 3)
Apparent total body clearance (CL/F) | Day 2 (Periods 1 and 2) and Day 6 (Period 3)
Apparent volume of distribution during the terminal elimination phase after oral (extravascular) administration (Vz/F). | Day 2 (Periods 1 and 2) and Day 6 (Period 3)

SECONDARY OUTCOMES:
Incidence of treatment-emergent AEs (including SAEs) categorized by severity and relationship to study drug. | 12 to 14 days after the last dose of study drug
  ECG, Clinical Laboratories, Vitals Signs and Physical Exams will be used as a safety measure to detect any AEs.

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, M.D., Study Director — Spero Therapeutics
Locations (1):
- Medical Facility, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No